CLINICAL TRIAL: NCT00095966
Title: A Phase II Study of BAY 43-9006/Gemcitabine for Advanced Pancreatic Cancer
Brief Title: Sorafenib and Gemcitabine in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02629; 13169B; CDR0000391850; NCI-6567; UCCRC-13169B; U01CA099118 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sorafenib; Gemcitabine

ARMS (1):
- Treatment (sorafenib tosylate and gemcitabine hydrochloride) (Experimental): Patients receive oral sorafenib twice daily on days 1-28 and gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
Sorafenib may stop the growth of tumor cells by stopping blood flow to the tumor and by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving sorafenib with gemcitabine may kill more tumor cells. This phase II trial is studying how well giving sorafenib together with gemcitabine works in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with locally advanced or metastatic adenocarcinoma of the pancreas treated with sorafenib and gemcitabine.

II. Determine the toxicity experienced by patients with advanced pancreatic cancer who are treated with sorafenib plus gemcitabine.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28 and gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced or metastatic disease

    * Locally advanced disease must extend outside the boundaries of a standard radiotherapy port
* Not amenable to curative surgery or radiotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Pleural effusion and ascites are not considered measurable lesions
  * Outside prior radiotherapy port
* No known brain metastases
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* More than 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis
* Bilirubin normal
* AST and/or ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or ongoing infection
* No other active malignancy
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to sorafenib or other study agents
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No prior antiangiogenic agents
* No prior cytotoxic chemotherapy for metastatic disease
* At least 4 weeks since prior adjuvant chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior gemcitabine
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior investigational drugs
* No prior sorafenib
* No prior MAPK signaling agents
* Concurrent warfarin anticoagulation allowed provided the following criteria are met:

  * Therapeutic on a stable warfarin dose
  * INR ≤ 3
  * Undergo weekly INR testing
  * No active bleeding or pathological condition that carries a high risk of bleeding
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-09; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST criteria | Up to 6 months

SECONDARY OUTCOMES:
Progression free survival | From start of treatment to progression or death, assessed up to 6 months
  Kaplan-Meier curves will be constructed.
Survival | At 6 months
  Specific attention will be given to the six-month survival rate, for which 90% confidence intervals will be generated.
Overall survival | Up to 6 months
  Kaplan-Meier curves will be constructed

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States